CLINICAL TRIAL: NCT04775147
Title: Intensive Control of Blood Pressure in Acute Ischemic Stroke After Endovascular Therapy on Clinical Outcome:A Prospective Multicenter Randomized Controlled Trial (CRISIS I)
Brief Title: Intensive Control of Blood Pressure in Acute Ischemic Stroke After Endovascular Therapy on Clinical Outcome (CRISIS I)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Results of ENCHANTED have been published.
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRISIS I
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2022-04

CONDITIONS: Acute Ischemic Stroke
Keywords: Mechanical thrombectomy; Blood pressure management
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Open intervention; outcome assessments undertaken by trained research staff who are kept blind to treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Achieving SBP level of <120mmHg within 1 hour after successful recanalization, and maintaining this level at least 72 hours.
  Interventions: Other: Intensive BP lowering
- Control group (No Intervention): Maintaining SBP level of <140mmHg within 1 hour after successful recanalization, and maintaining this level at least 72 hours.

INTERVENTIONS:
Other: Intensive BP lowering — The aim is to achieve a systolic BP level of <120mmHg within 1hour after successful recanalization and to maintain this BP level for the next 72 hours (or until hospital discharge or death of this should occur earlier)
  Arms: Intervention group

SUMMARY:
CRISIS I is a prospective, multicenter, randomized controlled trial, to asses the impact of intensive blood pressure control on clinical outcome of acute ischemic stroke patients with successful recanalization after endovascular therapy.

DETAILED DESCRIPTION:
CRISIS I aims to determine the effectiveness of more intensive BP lowering target (<120 mmHg) compared to standard BP management target (<140mmHg) on functional outcome in patients with successful recanalization post-MT for AIS due to anterior circulation large vessel occlusion (LVO).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of AIS with anterior circulation LVO confirmed by brain imaging
* To receive MT <24 hours after AIS onset according to local guidelines
* Successful recanalization (TICI score ≥2b) after MT
* Sustained systolic BP ≥140 mmHg (defined as 2 successive readings <10 mins) within 60 minutes after recanalization
* Provide written informed consent (or approved surrogate)
* Perform CTA or MRI before endovascular therapy
* Signed an approved informed consents

Exclusion Criteria:

* Significant pre-stroke disability (mRS scores 2-5)
* Definite indication/contraindication to different intensities of BP lowering treatment
* Specific contraindications to any of the BP agents to be used (eg, patients who are hypersensitive (allergic) to any of the ingredients)
* Unlikely to potentially benefit from therapy (e.g. advanced dementia) or very high likelihood of death within 24 hours post-MT, judged by responsible treating clinician
* Other medical illness that interferes with outcome assessments and follow-up (e.g.advance cancer and renal failure); Women who are lactating
* Other conditions inappropriate for inclusion judged by investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Level of disability | 90 days (3months)
  a shift (improvement) in scores (0-6) on the modified Rankin scale

SECONDARY OUTCOMES:
Intracerebral hemorrhage | 90 day
  Any or symptomatic ICH (sICH) after endovascular therapy
Death or neurological severity | 7 days
  Death or dependency measured by National Institutes of Health stroke scale (NIHSS)
BP lowering target (<120 mmHg) | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu, China